CLINICAL TRIAL: NCT06688721
Title: Does Eco-driving Assistance (EDA) Have an Impact on Bus Driver's Health and Well-being? A Pseudo-randomized Controlled Trial
Brief Title: Does Eco-driving Assistance (EDA) Have an Impact on Bus Driver's Health and Well-being?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2024-01573
Record Dates: First submitted 2024-11-01; First posted 2024-11-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Public transport; Eco-driving assistance; Occupational health; Health and well-being; Bus drivers

STUDY DESIGN:
Intervention Model Description: Within subject design Each participant will be allocated to both the intervention (i.e. driving shifts with EDA-equipped buses) and the control (i.e. driving shifts with non-EDA-equipped buses) conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDA (Experimental): Driving shifts with EDA-equipped buses
  Interventions: Device: Driving a bus equipped with EDA
- Control (No Intervention): Driving shifts with non-EDA-equipped buses

INTERVENTIONS:
Device: Driving a bus equipped with EDA — Eco-driving assistance (EDA) systems is a technology integrated into vehicles that helps drivers to optimize fuel efficiency and reduce emissions by providing real-time feedback and guidance on driving behaviors. The system typically analyzes several driving behaviours that are measured using different captors and sensors. These systems aim to reduce the overall carbon footprint of driving, leading to cost savings for the public transport company and reduced environmental impact.
  Arms: EDA

SUMMARY:
The goal of this pragamatic trial is to assess the impact of eco-driving assistance (EDA) system on professional bus drivers' health and well-being.

The main questions it aims to answer are:

* Does the eco-driving assistance (EDA) act as a stressor for bus drivers ?
* Does the physiological and psychological perceived stress increase when bus drivers are driving bus equipped with eco-driving assistance (EDA) ?

An additional question consists in assessing the association between stress measurements and biomarkers in biological samples.

Researchers will compare the heart rate variability (HRV) and perceived stress level when participant are allocated to EDA-equipped buses and non-EDA-equipped buses

Participants will:

* Drive buses equipped with eco-driving assistance (EDA)
* Drive buses without eco-driving assistance (EDA)
* Wear a wearable electrocardiogram (ECG) device (Bittium Faros) to record the heart rate variability (HRV)
* Answer a questionnaire at the end of each working day (end-of-service questionnaire)
* When allocated to bus with eco-driving assistance (EDA), read the EDA-generated report and answer some related questions in the end-of-service questionnaire
* Upon acceptance only, a collection of biological samples and physiological measurement will be performed

DETAILED DESCRIPTION:
This pragmatic pseudo-randomized trial will allow the investigators to assess the effect of eco-driving assistance (EDA) on bus drivers' health and well-being. Each bus driver will be randomly allocated to either buses equipped with eco-driving assistance (EDA) (i.e. intervention) and buses without eco-driving assistance (EDA) (i.e. control). The research team will use the within-subject design, allowing to allocate both the intervention and the control to each participant.

Throughout the working day, each bus driver will continuously wear an ECG device (Bittium Faros) to record the HRV. At the end of each working day, participants will receive a questionnaire (i.e. end-of-service questionnaire) to fill in. If they have been allocated to at least one EDA-equipped bus during their working day, they will need to read the EDA-generated report and come back to the questionnaire to fill in additionnal questions.

To record enough data, participants will need to reach at least 5 hours driving shifts with an EDA-equipped bus and 5 hours driving shifts without EDA. When this endpoint is reached, the study is over.

ELIGIBILITY:
Inclusion Criteria:

* adult active bus driver
* having signed the informed consent
* having worked for at least one year as TPF bus driver
* working at least 30 hours a week
* no planned extended absences in the next 6 months (civil service, military service, long- term leave, retirement)

Exclusion Criteria:

* wearing a medical active implant (pacemaker, cardiac defibrillator, neurostimulator, other electronic implant)
* known allergy or skin sensitivity to plasters

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | From enrollment in the study to at least 5 days and until the endpoint is reached (i.e. at least 5 hours driving shifts with buses equipped with EDA and 5 hours driving shifts with buses without EDA) but for a maximum duration of 14 days
  Heart rate variability (HRV) will be measured using the Bittium Faros ECG device. Participants will continuously wear the device throughout their working day and during one full non-working night, to obtain baseline value.

SECONDARY OUTCOMES:
Perceived stress | 1 day at the beginning of the study, once the eligibility has been confirmed
  Perceived stress will be assessed with the validated perceived stress scale questionnaire included in the baseline questionnaire, filled at the begining of the study, once the eligibility has been confirmed.
  For each question participants will choose from the following alternatives: 0 = never; 1 = almost never; 2 = sometimes; 3 = fairly often, 4 = very often
Perceived stress | From enrollment in the study to at least 5 days and until the endpoint is reached (i.e. at least 5 hours driving shifts with buses equipped with EDA and 5 hours driving shifts with buses without EDA) but for a maximum duration of 14 days
  Visual analog scale (VAS) for perceived stress during their working days included in the daily end-of-service questionnaire Scale from 0 to 100, with 0 = no stress and 100 = maximal stress
Perceived stress | From enrollment in the study to at least 5 days and until the endpoint is reached (i.e. at least 5 hours driving shifts with buses equipped with EDA and 5 hours driving shifts with buses without EDA) but for a maximum duration of 14 days
  Specific questions related to any stessful events encountered during the participant's working days included in the end-of-service questionnaire
Stress biomarkers in saliva samples | From enrollment in the study to at least 5 days and until the endpoint is reached (i.e. at least 5 hours driving shifts with buses equipped with EDA and 5 hours driving shifts with buses without EDA) but for a maximum duration of 14 days
  Saliva auto-collection (upon acceptance only) by participants to further measure cortisone and cortisol and correlate their levels with any participant reported stressful events in the end-of-service questionnaire.
Perceived stress linked with eco-driving assistance system generated report | From enrollment in the study to at least 5 days and until the endpoint is reached but for a maximum duration of 14 days and only when allocated to the intervention
  When allocated to the intervention (i.e. driving shifts with buses with eco-driving assistance), participants will need to read the EDA-generated report and answer few additional questions included the end-of-service questionnaire, including a visual analog scale (VAS) for the perceived stress while reading the report Scale from 0 to 100, with 0 = no stress and 100 = maximal stress

CONTACTS AND LOCATIONS:
Overall Officials: Irina Guseva Canu, Professor, Principal Investigator — Unisanté
Locations (1):
- TPF, Givisiez, Canton of Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All data generated during this study will be shared with restrictive access. Data are considered as coded as long as the identity of the participants involved is preserved.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available at the end of the project, once all the data have been collected
Access Criteria: IPD and supporting information (containing only coded data) will be stored on the secured institutional data repository (Unisanté repository).
  Access will be given upon request to the principal investigator.
URL: https://intranet.unisante.ch/document/871642/revision/895699

REFERENCES:
- [Derived] Krummenacher M, Ghosh M, Turner MC, Guseva Canu I. Protocol for a pseudo-randomized controlled trial to assess the impact of eco-driving assistance systems on bus drivers' stress responses. Environ Health Prev Med. 2025;30:90. doi: 10.1265/ehpm.25-00259. PMID 41242744